CLINICAL TRIAL: NCT02398539
Title: Randomized Clinical Trial Comparing Silver Nitrate Application With Topical Corticosteroids for Hypergranulation Tissue at Gastrostomy Sites
Brief Title: Silver Nitrate Application and Topical Corticosteroids for Hypergranulation Tissue
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Eloise Lemon, Principal Investigator, Akron Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150110
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Hypergranulation Tissue; Gastrostomy Tube Site
MeSH Terms: interventions — Silver Nitrate; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Silver nitrate treatment will include weekly applications in the pediatric surgery office by a clinician.
  Interventions: Drug: Silver Nitrate
- Group 2 (Active Comparator): Triamcinolone cream, 0.5% applied three times per day by the patient's caregiver.
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Silver Nitrate — Silver Nitrate Sticks
  Arms: Group 1
Drug: Triamcinolone — 0.5% cream
  Arms: Group 2

SUMMARY:
This protocol describes a randomized, two arm clinical trial comparing two topical treatments in patients with hypergranulation tissue at gastrostomy tube sites. The subjects are randomized to either group 1or group 2 treatments:

Maximum duration of therapy is 4 weeks. However, the therapy may be discontinued anytime at the discretion of the investigator or if there is resolution of the of the hypergranulation tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients <18
2. Evaluated for hypergranulation at the G-tube site
3. Inpatient and out-patient

Exclusion Criteria:

Children not meeting the above criteia

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Maximal reduction in granulation tissue | During maximum of 4 weeks of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States